CLINICAL TRIAL: NCT01341002
Title: Red Blood Cells (RBC) Transfusion Related to Central Venous O2 Saturation
Brief Title: Red Blood Cells (RBC) Transfusion Related to Central Venous O2 Saturation (ScvO2) Measurement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2008-A01247-48; 2008/0834 (Other: sponsor); B81159-60 (Other: AFSSAPS)
Record Dates: First submitted 2011-04-21; First posted 2011-04-25 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Postoperative Complications; Erythrocyte Transfusion; Oxygen Disorders
Keywords: Postoperative Care; red blood cell transfusion; venous oxygen saturation
MeSH Terms: conditions — Postoperative Complications | interventions — Blood Transfusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SCVO2 < 70% (Experimental): guidelines transfusion + SCVO2 < 70%
  Interventions: Procedure: Transfusion
- currently intervention (Active Comparator): guidelines transfusion
  Interventions: Procedure: Transfusion

INTERVENTIONS:
Procedure: Transfusion — Red Blood Cells (RBC) Transfusion if SCVO2 < 70% and guidelines
  Arms: SCVO2 < 70%
Procedure: Transfusion — transfusion based on guidelines
  Arms: currently intervention

SUMMARY:
The objective of this study is to estimate red blood cells (RBC) transfusion related to central venous O2 saturation (ScvO2) measurement. This prospective, randomized trial is performed in visceral, vascular and thoracic surgery units in the university hospital of Lille.

One hundred patients need to be included. Inclusion criteria are: age 18 to 99 year old, patient with central venous catheter in place and fulfilling the haemoglobin (Hb) threshold criteria for RBC transfusion according to the XXIIIth French Consensus Conference in critical care medicine recommendations.

After randomisation, patients will be eligible to receive RBC according to their level of Hb in the standard group and according to the Hb and ScvO2 in the optimization group. Patients without any disease are transfused if their Hb level is below 7g/dL; patients older than 60 years or having sepsis are transfused if their Hb level is 8g/dL or lower and cardiac patients are transfused if their Hb level is 9g/dL or lower. In the second group, transfusion is performed if and only if the ScvO2 level is les than 70% when Hb is under the same threshold levels.

The primary aim of the study is to compare the number of RBC units transfused by group (standard group or optimization group) over a period of 5 days counted from the first decision of transfusion taken post-operative. Considering the randomisation and considering the 50 % reduction of the decisions of transfusion in the group optimization, the absolute blood savings is estimated 25 % for the whole population. Secondary end points include the number of side effects associated with transfusion or when avoiding transfusion, length of hospital stay, and hospital mortality as well as major adverse events.

DETAILED DESCRIPTION:
red blood cells central venous O2 saturation surgery transfusion XXIIIth French Consensus Conference adult

ELIGIBILITY:
Inclusion Criteria:

* central venous catheter
* anemia With reference to french consensus about transfusion

Exclusion Criteria:

* intensive care
* emergency transfusion
* shock, hypovolemia
* need to go under surgery into 4 hours
* acute kidney injury or chronic renal disease
* brain injury
* pregnancy
* heart disease : ischemia <1 mois

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-11; Primary Completion 2013-11 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Number of RBC units transfused by group | 5 days
  to compare the number of RBC units transfused by group (standard group or optimization group) over a period of 5 days counted from the first decision of transfusion taken post-operative

CONTACTS AND LOCATIONS:
Overall Officials: Benoît VALLET, PU-PH, Principal Investigator — Lille University Hospital
Locations (1):
- university Hospital, lille, Lille, France